CLINICAL TRIAL: NCT02523040
Title: A Phase II Study of Lenalidomide for Adult Histiocyte Disorders
Brief Title: Lenalidomide for Adult Histiocyte Disorders
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, Eric Jacobsen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-197
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Results first posted 2025-04-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Langerhans Cell Histiocytosis (LCH); Histiocytoses Erdheim-chester Disease; Histiocytic Sarcoma (HS)
Keywords: Langerhans cell histiocytosis (LCH); Erdheim-Chester disease (ECD); Histiocytic Sarcoma (HS)
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Histiocytic Sarcoma; Erdheim-Chester Disease | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): After the screening procedures confirm participation in the research study.
  - Lenalidomide Oral, Daily for 21 days of each cycle
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid

SUMMARY:
This research study is studying a chemotherapy drug Lenalidomide as a possible treatment for one of three histiocyte disorders: Langerhans cell histiocytosis (LCH), Erdheim-Chester disease (ECD), or histiocytic sarcoma (HS).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved lenalidomide for your specific disease but it has been approved for other uses. Lenalidomide is a chemotherapy drug that belongs to a class of drugs called immunomodulatory drugs (IMiDs), which modify a participant's immune response in order to treat cancer. Lenalidomide alters the body's immune system and it may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, it may reduce or prevent the growth of cancer cells. Lenalidomide has been shown to restore the immune cells' ability to attack and kill tumor cells Lenalidomide is approved by the FDA to treat certain cancers including multiple myeloma and myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed LCH, ECD or HS. Confirmation of outside pathology at BWH will be performed but is not mandatory prior to study enrollment (see section 3).
* Detectable disease by at least one of the following modalities: CT, PET, bone scan, or MRI.
* Patients with LCH must require systemic therapy according to the Histiocyte Society LCH Evaluation and Treatment Guidelines (HS 2009)

  -- Or
* Patients with HS requiring systemic treatment as defined by disease that cannot be surgically resected and/or encompassed in a single radiation field.
* Age 18 years or older.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within 1.5 times normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional upper limit of normal
  * creatinine within 2 times normal institutional limits

    --- OR
  * creatinine clearance ≥30 mL/min/1.73 m2. Note, dose adjustments are required for CrCl ≥30 mL/min but ≤60 ml/min.
* Able to take aspirin 81 mg daily as prophylactic anticoagulation if not on warfarin, low molecular weight heparin or oral factor Xa inhibitor. Patients intolerant to ASA may use warfarin or low molecular weight heparin at doses designed to treat deep venous thrombosis.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior chemotherapy or radiation within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Participants who are receiving any other investigational agents.
* Prior treatment with lenalidomide. Patients previously treated with thalidomide who discontinued treatment for reasons aside from an adverse reaction to thalidomide are permitted.
* History of another invasive malignancy unless treated with curative intent 5 years or more prior to study entry. Patients with localized carcinoma of the cervix, non-melanoma skin cancer, or early stage prostate cancer requiring observation only are eligible regardless of timing of diagnosis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because lenalidomide has known teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with lenalidomide, breastfeeding should be discontinued if the mother is treated with lenalidomide.
* Known active hepatitis B (HBV) or hepatitis C (HCV) infection. Patients who are positive only for HBV surface antibody as a result of prior vaccination are eligible. Patients with a positive HBV core antibody but undetectable HBV viral load are eligible.
* HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with lenalidomide. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Concomitant corticosteroids unless patient has been on a stable dose of prednisone (or equivalent) of ≤10 mg daily for at least 2 weeks prior to first dose of study drug.
* Inability to swallow pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2024-02 (Actual); Study Completion 2026-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jacobsen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: Single agent lenalidomide (len) orally days 1-21 of a 28-day cycle up to 12 cycles. During cycle 1 patients receive 10mg len. If tolerated well, dose increases to 25mg and, if not, dose is reduced to 5mg. Dose also dependent on creatinine clearance (CrCl) level. For patients not already receiving systemic anticoagulation, a minimum aspirin dose of 81mg daily or for one month following treatment discontinuation is required.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 12
Evaluable for TNF-Alpha Evaluable for TNF Alpha (Participants with baseline and at least one on-treatment cycle TNF-alpha measurement.) | 6
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 44 [23 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
ECOG performance status [Count of Participants; unit: Participants]
  00 - Fully Active | 4
  01 - Restricted | 7
  02 - Ambulatory and Capable of Self Care | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Proportion of participants achieving either complete resolution of all signs or symptoms which is non-active disease (NAD) status or regression of signs or symptoms along with no new lesions which is better active-disease (AD) status per Histiocyte Society criteria any time on treatment.
Time Frame: Disease assessed every 3 cycles on treatment up do 12 cycles (approximately 12 months).
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
proportion of participants | 0.67 [0.39 to 0.88]

2. Secondary Outcome: 12-months Progression-free Survival (PFS)
Description: Progression-free survival (PFS) based on the Kaplan-Meier method is defined as time from registration to progression (PD) or death, censored for patients alive and progression-free at last disease assessment. PD is defined by Histiocyte criteria. Percent PFS is the percent of patients who are alive and progression-free at 12 months.
Time Frame: Disease assessed on treatment every 3 cycles and in long-term follow-up up to the earlier of 36 months (every 3 months for 2 years then every 6 months) or start of new anti-cancer therapy. Relevant for this endpoint was12-months estimate.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
percentage probability | 62 [39 to 100]

3. Secondary Outcome: 12-months Overall Survival (OS)
Description: Overall survival (OS) based on the Kaplan-Meier method is defined as the time from registration to death, censored for patients alive at last contact. Percent OS is the percent of patients who are alive at 12 months.
Time Frame: 12 Months
Population: Survival followed up 36 months from start of protocol treatment. Relevant for this endpoint was12-months estimate.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
percentage probability | 92 [77 to 100]

4. Secondary Outcome: Incidence of Grade 3-4 Toxicity
Description: Grade 3-4 adverse events (AE) with treatment attribution of possibly, probably or definite (treatment-related) based on NCI Common Toxicity Criteria for Adverse Events version 3 (CTCAEv3) as reported on case report forms were tabulated by maximum grade. Incidence is the proportion of participants experiencing at least one treatment-related grade 3-4 AE of any type during the time of observation.
Time Frame: Up to 12 months on treatment.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Groups:
- Lenalidomide: After the screening procedures confirm participation in the research study.
  - Lenalidomide Oral, Daily for 21 days of each cycle
  Lenalidomide
Arm/Group | Lenalidomide
Number analyzed (Participants) | 12
proportion of participants | 0.25 [0.07 to 0.53]

5. Secondary Outcome: Urine Cell Free DNA for BRAF
Description: Quantitative serial measurements of urine cell free DNA for BRAF mutation as a biomarker of response
Time Frame: 12 Months
Reporting Status: Not Posted

6. Secondary Outcome: Percent Change in Serum TNF-alpha Levels on Therapy From Baseline up to 12 Cycles
Description: Serum TNF-alpha levels were quantified per established methods and maximum percent change in level from baseline derived.
Time Frame: Measured at baseline, day 1 of cycles 3, 6 ad 12 cycles and within 28 days post-treatment end (up to 13 months).
Population: Participants with baseline and at least one on-treatment cycle TNF-alpha measurement.
Measure: Median (Full Range); unit: percent change from baseline
Arm/Group | Lenalidomide
Number analyzed (Participants) | 6
percent change from baseline | -14.4 [-67.3 to 8.3]

7. Secondary Outcome: Plasma Cell Free DNA for BRAF
Description: Quantitative serial measurements of plasma cell free DNA for BRAF mutation as a biomarker of response
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=12)
Fatigue (General disorders) | 10 (12)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (19)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Neutrophil count decreased (Investigations) | 5 (16)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (5)
Headache (Nervous system disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (6)
Platelet count decreased (Investigations) | 4 (6)
Dizziness (Nervous system disorders) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema limbs (General disorders) | 3 (3)
White blood cell decreased (Investigations) | 3 (6)
Alanine aminotransferase increased (Investigations) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Edema face (General disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Bilateral orbital lesions
Eye pain (Eye disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) — Facial asymmetry Rhinorrhea
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Polydipsia
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle cramps
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Mental haziness
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Weight gain (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT02523040/Prot_SAP_000.pdf